CLINICAL TRIAL: NCT06167577
Title: Dysbindin-antipsychotics Psychophamarcogenetics: a Mouse-human Translational Study Towards Personalized Healthcare in Bipolar Disorders GR-2016-02362413
Brief Title: Dysbindin-antipsychotics Psychophamarcogenetics: a Mouse-human Translational Study Towards Personalized Healthcare in Bipolar Disorders
Acronym: DYSBIP
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: ASST Santi Paolo e Carlo (Other); Asst Melegnano e Martesana (Other Government); Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: DYSBIP
Record Dates: First submitted 2023-11-10; First posted 2023-12-12 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2022-11

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; disbindina; antipsychotic
MeSH Terms: conditions — Bipolar Disorder | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Psychometric scales (BPRS, MRS, HAM-D, SES, and GAF) monthly — we will correlate the clinical/neuropsychological response to antipsychotics with the presence of the functional DysBray haplotype of the DTNBP1 gene
  Other Names: A single blood sample collection at study entry (T0) for the genotyping of the DTNBP1 gene (functional DysBray haplotype).

SUMMARY:
We will conduct an observational study involving a preliminary long-term follow-up designed to test how dysbindin-1 gene expression can modulate the efficacy of treatments with antipsychotics on clinical and neuropsychological outcomes. We will recruit 150 patients diagnosed with DB who required therapy with an atypical antipsychotic (aripiprazole or quetiapine or olanzapine) in combination with a medication mood stabilizer (lithium or other mood stabilizer), according to the standards of DB treatment. Treatment will be maintained stably for at least 6 months, unless the patient's clinical evolution makes a therapeutic switch inevitable. In light of the data in mice, we will correlate the clinical/neuropsychological response to antipsychotics with the presence of the functional DysBray haplotype of the DTNBP-1 gene, which has in the general population a relatively high prevalence (about 25 percent).

DETAILED DESCRIPTION:
During the first visit, all subjects will sign informed consent and undergo a a clinical interview, in which clinical data will be collected. The demographic information will be transcribed into the electronic data collection form ("Electronic case report forms" - eCFR). The electronic data collection form should be completed at the time of the visit, so that it can objectively report the most recent observations. Each month recruited subjects will be administered specific scales (BPRS, YMRS, HAM-D, SES, GAF) validated in order to assess the psychopathological component. In addition, at the beginning of the study, a neuropsychological evaluation will be conducted to assess the cognitive status of the recruited patients. Therefore, neuropsychological tests will be administered. standardized (WAIS, BAC-A). In addition, neuropsychological assessments will be carried out as a follow-up (administration of the BAC-A) every 6 months, culminating in a follow-up of at least 12 months, to monitor the cognitive status of the subjects. Information obtained during the conduct of this clinical study is confidential and disclosure to third parties other than those indicated is strictly prohibited. The data collected (all information contained in original documents and certified copies or results clinical trials, observations or other activities in a clinical trial necessary for the reconstruction and evaluation of the study) will be archived in the file. The documents will be stored in a specific locked filing cabinet. The information collected will then be entered into a database, a management system (e.g., Microsoft Access). The data will be constantly backed up at the end of each week to prevent the loss of data that have been stored on the server. A server failure will cause delays in the execution phase of the analyses. The investigator must maintain all study records according to the guidelines on Good Clinical Practice (CGP) "International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH)" and according to the record retention policies of the country in which the study. In accordance with the ICH/GCP guidelines, the investigator/institution will maintain all electronic resources and all original documents that support the data collected from each subject and all study documents (documents essential to the conduct of a study clinical trial). The investigator/institution will take measures to prevent the destruction accidental or premature destruction of these documents. Essential documents must be kept for at least 2 years after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* DB diagnoses, made by the use of the structured clinical interview based on the DSM-5 criteria (SCID-CV);
* Therapy with an atypical antipsychotic (aripiprazole or quetiapine or olanzapine) in combination with a mood stabilizer (lithium or another mood stabilizer mood), according to the standard of care.

Exclusion Criteria:

* Comorbidity with other psychiatric disorders;
* comorbidity with neurological disorders, with damage to the brain and with deficits intellectual;
* pregnancy;
* current and past substance abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bipolar disease patients who required therapy with an atypical antipsychotic in combination with a mood stabilizer
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
analyze the impact of genetic variants of the Disbindin-1 gene on patient's response to antipsychotic drugs | 12 months
  Patients will undergo a follow-up lasting at least 12 months, during which we will we will record: Number and duration of illness relapses (hypomanic/manic, mixed or depressive), the number of emergency room admissions, hospitalizations, attempted suicide; Assessment of clinical and psychopathological status by psychometric scales (BPRS, MRS, HAM-D, SES and GAF) every month; Assessment of cognitive status through neuropsychological tests standardized (WAIS, BAC-A) every 6 months; A single blood sample collection at study entry (TO) for the DTNBP1 gene genotyping (DysBray functional haplotype (12).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grande I, Berk M, Birmaher B, Vieta E. Bipolar disorder. Lancet. 2016 Apr 9;387(10027):1561-1572. doi: 10.1016/S0140-6736(15)00241-X. Epub 2015 Sep 18. PMID 26388529
- [Background] Merikangas, K.R., et al. Archives of general psychiatry 68, 241-251 (2011).
- [Background] Hasan A, Falkai P, Wobrock T, Lieberman J, Glenthoj B, Gattaz WF, Thibaut F, Moller HJ; WFSBP Task force on Treatment Guidelines for Schizophrenia. World Federation of Societies of Biological Psychiatry (WFSBP) guidelines for biological treatment of schizophrenia, part 2: update 2012 on the long-term treatment of schizophrenia and management of antipsychotic-induced side effects. World J Biol Psychiatry. 2013 Feb;14(1):2-44. doi: 10.3109/15622975.2012.739708. Epub 2012 Dec 6. PMID 23216388
- [Background] Ji, Y., et al. Proceedings of the National Academy of Sciences of the United States of America 106,19593-19598 (2009).
- [Background] Li W, Zhang Q, Oiso N, Novak EK, Gautam R, O'Brien EP, Tinsley CL, Blake DJ, Spritz RA, Copeland NG, Jenkins NA, Amato D, Roe BA, Starcevic M, Dell'Angelica EC, Elliott RW, Mishra V, Kingsmore SF, Paylor RE, Swank RT. Hermansky-Pudlak syndrome type 7 (HPS-7) results from mutant dysbindin, a member of the biogenesis of lysosome-related organelles complex 1 (BLOC-1). Nat Genet. 2003 Sep;35(1):84-9. doi: 10.1038/ng1229. Epub 2003 Aug 17. PMID 12923531
- [Background] Talbot K, Cho DS, Ong WY, Benson MA, Han LY, Kazi HA, Kamins J, Hahn CG, Blake DJ, Arnold SE. Dysbindin-1 is a synaptic and microtubular protein that binds brain snapin. Hum Mol Genet. 2006 Oct 15;15(20):3041-54. doi: 10.1093/hmg/ddl246. Epub 2006 Sep 15. PMID 16980328
- [Background] Papaleo F, Yang F, Garcia S, Chen J, Lu B, Crawley JN, Weinberger DR. Dysbindin-1 modulates prefrontal cortical activity and schizophrenia-like behaviors via dopamine/D2 pathways. Mol Psychiatry. 2012 Jan;17(1):85-98. doi: 10.1038/mp.2010.106. Epub 2010 Oct 19. PMID 20956979
- [Background] Papaleo, F., Burdick, M.C., Callicott, J.H. & Weinberger, D.R. Mol Psychiatry 19, 311- 316(2014). 12. Bray, N.J.,et al. Hum Mol Genet 14, 1947-1954 (2005).
- [Background] Boscutti A, Pigoni A, Delvecchio G, Lazzaretti M, Mandolini GM, Girardi P, Ferro A, Sala M, Abbiati V, Cappucciati M, Bellani M, Perlini C, Rossetti MG, Balestrieri M, Damante G, Bonivento C, Rossi R, Finos L, Serretti A, Brambilla P, The Gecobip Group. The Influence of 5-HTTLPR, BDNF Rs6265 and COMT Rs4680 Polymorphisms on Impulsivity in Bipolar Disorder: The Role of Gender. Genes (Basel). 2022 Mar 9;13(3):482. doi: 10.3390/genes13030482. PMID 35328036